CLINICAL TRIAL: NCT06862895
Title: Effect of Chest Physiotherapy Educational Program on Mother's Knowledge, Practice and Clinical Outcomes of Infants With Bronchiolitis
Brief Title: Effect of Chest Physiotherapy on Clinical Outcome of Infants With Bronchiolitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Shaimaa Shwan, principal Investigator, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CPT
Record Dates: First submitted 2025-01-29; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Bronchiolitis; Infant, Newborn, Diseases; Chest Physiotherapy; Educational Program
MeSH Terms: conditions — Bronchiolitis; Infant, Newborn, Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): chest physiotherapy
  Interventions: Other: chest physiotherapy
- control group (No Intervention): no intervention

INTERVENTIONS:
Other: chest physiotherapy — Chest Physiotherapy is including various techniques, in this study classical CPT was used to be applied to participants
  Arms: intervention group

SUMMARY:
The goal of clinical trial study is to evaluate effect of chest physiotherapy educational on mother's knowledge, practice and clinical outcomes of infants aged less than 12 months diagnosed with bronchiolitis by physician

The main questions aims to answer:

* Does chest physiotherapy improve clinical outcomes of infants with bronchiolitis?
* Does educational program improve mothers knowledge and practice regarding chest physiotherapy?

Researcher compare two groups one receive routine hospital care (control group) other receive chest physiotherapy applied by mothers in addition to routine hospital care and will be followed up for 3 days

ELIGIBILITY:
Inclusion Criteria:

* 1. Mothers of infants diagnosed with bronchiolitis. 2. Presence of crackle on auscultation.

Exclusion Criteria:

1. Children with contraindication of chest physiotherapy (ex. Fracture, recent surgery)
2. Children who intubated and admitted to Intensive Care Unit (ICU).

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
change in Clinical Outcomes of Infants with Bronchiolitis | baseline
  changing of oxygen saturation( SPO2) <90% to normal level SPO2>92%
change in physiological outcomes of Infants with Bronchiolitis | baseline
  change in respiratory rate from abnormal to normal (0-3 month RR:35-55 3-6 month RR:30-45 6-12 month RR:25-40) breath per minute

SECONDARY OUTCOMES:
Improvement in Knowledge of Mother's | After 3 days
  after application of educational program expected to to improve mother's knowledge regarding chest physiotherapy
Improvement in practices of Mother's | After 3 days
  after application of educational program expected to to improve mother's practice regarding chest physiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Hawler Medical University, Erbil, Kurdistan, Iraq

IPD SHARING:
Plan to Share IPD: No